CLINICAL TRIAL: NCT02006316
Title: Beneficial Effects of Microsurgical Varicocelectomy on Semen Parameters in Patients Who Underwent Surgery for Causes Other Than Infertility
Brief Title: Beneficial Effects of Microsurgical Varicocelectomy on Semen Parameters for Causes Other Than Infertility
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo Woong Kim, MD, Professor, Seoul National University Hospital
Other Study IDs: SeoulNUH
Record Dates: First submitted 2010-03-17; First posted 2013-12-10 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- varicoceles: men with clinical varicoceles underwent microsurgical varicocelectomy due to causes other than infertility such as testicular pain, discomfort or scrotal mass
  Interventions: Procedure: Microsurgical subinguinal varicocelectomy

INTERVENTIONS:
Procedure: Microsurgical subinguinal varicocelectomy

SUMMARY:
The purpose of this study is to evaluate whether clinical varicoceles are associated with abnormal semen parameters and whether varicocelectomy could improve the semen parameter in patients unrelated with infertility.

DETAILED DESCRIPTION:
While most studies are continued to validate the observations of significant improvements in sperm density and motility after varicocele ligation in infertile patients, there have been few studies to investigate the effects of varicocelectomy on semen parameters in adult men unrelated with infertility. The purpose of this study was to determine whether varicocelectomy could improve the semen parameter of these patients as well as whether clinical varicoceles are associated with abnormal semen parameters in patients unrelated with infertility.

ELIGIBILITY:
Inclusion Criteria:

* men with clinical varicoceles underwent microsurgical varicocelectomy due to causes other than infertility such as testicular pain, discomfort or scrotal mass

Exclusion Criteria:

* adolescents
* men with proven fertility or azoospermia
* men with preoperative normal sperm analysis
* available data to compare between preoperative and postoperative semen analyses

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: men with clinical varicoceles underwent microsurgical varicocelectomy due to causes other than infertility such as testicular pain, discomfort or scrotal mass
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2000-01; Primary Completion 2008-04 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sperm concentration, motility, and morphology | at postoperative 4months
  To observe the change of sperm concentration, motility, and morphology pre and postoperatively in the patients of inclusion criteria

SECONDARY OUTCOMES:
whether semen analysis should be done in men with clinical varicocele regardless of the chief complaint | at postoperative 4months
  this result would show the need of performing semen analysis even in the patients with clinical varicocels due to causes other than infertility

CONTACTS AND LOCATIONS:
Overall Officials: Soo Woong Kim, M.D.,Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea